CLINICAL TRIAL: NCT04505072
Title: Randomized Controlled Study of PR-ESSENCE - a Problem Solving Model for Youth With Challenging Behavior in Special (SiS) Treatment Homes
Brief Title: RCT of PR-ESSENCE - a Problem Solving Model for Youth With Challenging Behavior in Special (SiS) Treatment Homes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GNC SiS PR-ESSENCE
Record Dates: First submitted 2020-08-02; First posted 2020-08-07 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Behavior Problems; Neurodevelopmental Disorders
MeSH Terms: conditions — Mental Disorders; Neurodevelopmental Disorders | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Primary outcome assessed by blinded rater
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PR-ESSENCE treatment (Experimental): PR-ESSENCE treatment 10 weeks
  Interventions: Behavioral: PR-ESSENCE
- Control (Active Comparator): Treatment as usual 10 weeks
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: PR-ESSENCE — Manual-based training of mutual problem-solving
  Arms: PR-ESSENCE treatment
Behavioral: Treatment as usual — General support in daily structure and activities that is given to all youth staying at the treatment homes
  Arms: Control

SUMMARY:
Randomized controlled trial of PR-ESSENCE treatment for youth with challenging behavior in two youth treatment homes, including 60-70 youth. Inclusion criteria: Youth aged 12-17 years, staying at least 3 months at the home, with intellectual function in the normal range according to WISC-test and clinical judgment, and exhibiting significant problem behaviors as measured by Broset Violence Checklist (BVC). Subjects are randomized to 10 weeks of PR-ESSENCE treatment or to the control condition "treatment as usual". After the control period, the control group will receive 10 weeks of PR-ESSENCE treatment. Outcome is assessed at baseline, post-treatment/control period, and 3-6 months post-treatment (at the time when the youth is planned to move from the home) with global assessments of problem severity and improvement by blinded rater (CGI-I, CGI-S), ratings of SNAP-IV (ADHD and oppositional symptoms), ECBI (behavior problems) and RPQ (relation problems) by the youth's contact person, and self-ratings of psychiatric symptoms and self-concept with Becks Youth Inventories. BVC ratings are also made daily by contact persons and teachers during the whole study.

DETAILED DESCRIPTION:
PR-ESSENCE is a problem-solving training program developed by our research team, inspired by Dr Greene´s model "Collaborative and Proactive Solutions (CPS)". We recently completed an RCT with PR-ESSENCE at the Gillberg Centre, Gothenburg University, including 108 children and adolescents who had complex neurodevelopmental disorders such as autism, ADHD, ODD, Tourette, learning difficulties etc and challenging behaviors. The study showed significant global improvements in behavior problems with a large effect size.

The PR-ESSENCE model is designed to train and develop mutual problem solving strategies for children and adolescents with neurodevelopmental disorders (ESSENCE, an umbrella term coined by Gillberg 2010 = Early Symptomatic Syndromes Eliciting Neuropsychiatric Clinical Examinations, which puts focus on the considerable overlap several of these syndromes have). Many youth who are placed in youth treatment homes due to challenging and risk-taking behaviors have been shown to have ESSENCE impairments.

The present study is a randomized controlled trial of PR-ESSENCE treatment for youth with challenging behavior in two youth treatment homes in southwestern Sweden, Bjorkbacken (girls) and Nereby (boys). We plan to include 60-70 youth. Inclusion criteria: Youth aged 12-17 years, staying at least 3 months at the home, with intellectual function in the normal range according to WISC-test and clinical judgment, and exhibiting significant problem behaviors as measured by Broset Violence Checklist (BVC). Exclusion criteria: Intellectual disability, bipolar syndrome, psychosis, substance use, or other unstable psychiatric or medical condition which would make study participation unsuitable. Psychoactive medication is allowed if stable at least one month before baseline, and during the trial.

At baseline a medical and neuropsychiatric history is taken by psychologist and physician (a standard assessment done for all youth placed at the homes), including rating of history of risk behaviors with Youth Level of Service/Case Management Inventory (YLS/CMI), and a DSM-5-diagnostic screening (DSM-5-CCSM) for psychiatric symptoms. Intellectual level will be tested with WISC-V. The participants will do self-ratings of psychiatric symptoms and self-concept with Becks Youth Inventories. The therapists interview parents/carers about history of neuropsychiatric symptoms with the A-TAC-interview.

Subjects are randomized to 10 weeks of PR-ESSENCE treatment or to the control condition "treatment as usual". After the control period, the control group will also receive 10 weeks of PR-ESSENCE treatment. Outcome is assessed at baseline, post treatment/control period, and 3-6 months post-treatment (at the time when the youth is planned to move from the home) with global assessments of problem severity and improvement by blinded independent rater (CGI-I, CGI-S), ratings of SNAP-IV (ADHD and oppositional symptoms), ECBI (behavior problems) and RPQ (relation problems) by the youth's contact person, and self-ratings of psychiatric symptoms and self-concept with Becks Youth Inventories. BVC ratings are made daily by contact persons and teachers during the whole study. During treatment, therapists rate every week with a Problem Rating Scale how many problem situations are completely or partly solved.

ELIGIBILITY:
Inclusion Criteria:

1. Youth with problem behaviors, placed for at least 3 months in the youth treatment homes Nereby (boys) and Bjorkbacken (girls).
2. Age 12-17 years
3. Intellectual function in the normal range according to WISC-test and clinical judgment
4. Problem behavior score of at least 5 points in one week on the Broset Violence Checklist (BVC). Score is measured during 2 weeks before screening
5. Medium to high-risk score on the YLS/CMI behavior problem domain 7
6. Psychotropic medication is allowed if stable during one month before baseline and during the randomized period of the trial

Exclusion Criteria:

1. Intellectual disability, bipolar syndrome, psychosis, substance use, or other unstable psychiatric or medical condition that would make study participation unsuitable

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2021-02-10 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression- Improvement (CGI-I) | 10 weeks, change
  Global rating of improvement by blinded rater based on all available information, score range 1-7, lower is better

SECONDARY OUTCOMES:
Clinical Global Impression- Severity (CGI-S) | 10 weeks, change
  Global rating of symptom severity by blinded rater based on all available information, score range 1-7, lower is better
Broset Violence Checklist (BVC) | 10 weeks, change
  Measures problem behaviors frequency/intensity, score range 0-36 per day, lower is better
SNAP-IV | 10 weeks, change
  Measures ADHD and Oppositional Defiant symptoms, score range ADHD 0-54, ODD 24, lower is better
Eyberg Child Behavior Inventory (ECBI) | 10 weeks, change
  Measures behavior problems frequency/intensity, score range 36-252, lower is better
Relationship Problems Questionnaire (RPQ) | 10 weeks, change
  Measures relationship problems, score range 0-30, lower is better

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Gillberg, Professor, Study Chair — Gillberg Neuropsychiatry Centre, Gothenburg University
Locations (1):
- Gillberg Neuropsychiatry Centre, Gothenburg, V. Gotaland, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04505072/Prot_SAP_000.pdf